CLINICAL TRIAL: NCT05646407
Title: Move With Air: Can a Fan Maximize the Benefits of a Supervised Exercise-training Program in Adults With Cardiopulmonary Disease?
Brief Title: Move With Air: Exercise Training Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Dennis Jensen, Ph.D., Associate Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FanEx 2023-9286
Record Dates: First submitted 2022-12-05; First posted 2022-12-12 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Chronic Obstructive Pulmonary Disease; Interstitial Lung Disease; Heart Failure
Keywords: Breathlessness; Dyspnea; Exercise; Fan-to-face therapy; Cool air; Exercise intolerance
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial; Heart Failure; Dyspnea; Motor Activity

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant
Masking Description: It is impossible to blind the participants or the investigators for the intervention, as they will be able to see whether they have been allocated to the fan-to-face group or the no fan group. However, participants will complete the supervised exercise-training sessions alone (with the study coordinator) with no other participants in the room, therefore they will be unaware of who has been allocated to the fan-to-face group or the no fan group. They will also be kept relatively unaware of the study hypothesis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise training with Fan-to-face (Experimental): Participants randomized to the fan-to-face group will perform supervised exercise training with a basic, portable fan (Honeywell HT-900 Turbo Force Air Circulator). The fan will be placed to the front of the treadmill with airflow directed toward the area of the face innervated by the second and third branches of the trigeminal nerve. The airflow speed will be chosen by each participant so that it is most comfortable to them. An anemometer will measure the airflow from the fan.
  Interventions: Device: Honeywell HT-900 Turbo Force Air Circulator
- Exercise training with no fan (No Intervention): Participants randomized to the no fan group will perform supervised exercise training with no fan. The exercise duration and intensity titration will follow the same format as the experimental group.

INTERVENTIONS:
Device: Honeywell HT-900 Turbo Force Air Circulator — This is a basic, portable, household fan with a single cost of CDN$21.99.
  Other Names: Fan
  Arms: Exercise training with Fan-to-face

SUMMARY:
The purpose of this study is to explore the role of a stream of cool air to the face, through fan-to-face therapy, as a novel adjunct non-pharmacological therapy to enable symptomatic adults with cardiopulmonary disease to exercise at higher intensities for longer durations and maximize the psycho-physiological benefits of a supervised exercise training program. The investigators hypothesize that, compared to no fan, fan-to-face therapy will result in relatively greater improvements in exercise endurance time and intensity ratings of perceived breathlessness during constant-load cardiopulmonary exercise testing on a treadmill at 75% of peak power output following a 5-week exercise training period.

DETAILED DESCRIPTION:
Prospective participants will complete four assessment visits (V1-V4) and 15 supervised exercise-training (T1-T15) sessions (3 sessions per week for 5 weeks). The purpose of visit 1 (V1) is twofold: 1) to screen potential participants for study eligibility; and 2) for participants identified as eligible, complete pulmonary function testing and an incremental exercise treadmill test to determine the relative intensity for visit 2 (V2). At V2, participants will undergo a dual-energy x-ray absorptiometry (DEXA) scan to assess body composition prior to the 5-week supervised exercise training. Participants will also perform an exercise endurance treadmill test at V2 performed at 75% of peak power achieved on the incremental exercise test from V1. Following V2, participants will be randomized to 5-weeks of 3x/week (total of 15 sessions) supervised exercise training to one of the two experimental conditions: (i) fan-to-face; or (ii) no fan (control). Exercise sessions will be individualized based on participants' ITT and progressed to ensure the participant is exercising at an intensity corresponding to a breathlessness intensity rating of between 3-5 Borg CR10 units and can complete at least 10 to 20-min of continuous walking. Exercise duration will be increased in 1 to 5-min intervals up to a maximum of 40-min. Thereafter, exercise intensity will be increased by 5-15% of baseline speed. Visit 3 (V3) will be done after the completion of the 5-week exercise training and will comprise of a second DEXA scan to assess for changes in body composition and the same exercise endurance test at V2 to assess for changes in exercise endurance time. Visit 4 (V4) will comprise of the same incremental exercise test as V1 to assess for changes in cardiovascular fitness.

ELIGIBILITY:
Inclusion Criteria:

* have a physician diagnosis of cardiopulmonary disease (e.g., chronic obstructive pulmonary disease, interstitial lung disease, heart failure)
* have a body mass index of >18.5 kg/m2 and <35 kg/m2
* be cleared to participate in a supervised exercise training program by their primary care physician

Exclusion Criteria:

* have changed their respiratory or cardiac medication dosage and/or frequency of administration in preceding two weeks
* have had a disease exacerbation/hospitalization in preceding six weeks
* have important contraindication(s) to exercise (e.g., significant musculoskeletal or neurological disease) or pulmonary function testing (e.g., eye, chest or stomach surgery, or any history of coughing up significant amounts of blood in the previous 3 months).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Cardiopulmonary exercise testing endurance time | Pre- and post-5 week of exercise training period.
  Cardiopulmonary exercise testing (constant-load at 75% peak power output) will be used to assess changes in endurance time pre to post intervention. Endurance time will be defined as the total duration of loaded walking (minutes).
Borg modified 0-10 category ratio scale for breathlessness intensity | Pre- and post-5 week of exercise training period.
  Borg modified 0-10 category ratio scale will be used to assess breathlessness intensity during constant-load (75% peak power output) cardiopulmonary exercise test at iso-time, defined as the highest equivalent 2-min interval of exercise completed by a given participant during each of the constant-load cardiopulmonary exercise test. A higher score is indicative of greater breathlessness, while a lower score is indicative of lesser breathlessness.

SECONDARY OUTCOMES:
Dual-Energy X-Ray Absorptiometry-derived body composition | Pre- and post-5 week of exercise training period.
  Dual-Energy X-Ray Absorptiometry will be used to assess changes in fat free mass pre to post supervised exercise training program. Fat free mass will be expressed as fat free max index, which is fat free mass per kg of total body weight per metre squared of standard height.
Cardiopulmonary exercise test physiological response (gas exchange) | Pre- and post-5 week of exercise training period.
  Breath-by-breath cardiopulmonary exercise test (incremental) parameters will be averaged in 30-second intervals at rest and during exercise. The change in peak volume of oxygen consumption pre to post supervised exercise training will be reported.
  A greater volume of oxygen consumption is indicative of a greater cardiovascular fitness
Cardiopulmonary exercise test physiological response (power output) | Pre- and post-5 week of exercise training period.
  Breath-by-breath cardiopulmonary exercise test (incremental) parameters will be averaged in 30-sec intervals at rest and during exercise. The change in peak power output pre to post supervised exercise training will be reported. A greater peak power output is indicative of greater leg strength and indirectly, cardiovascular fitness.
Minimal clinically important difference breathlessness intensity | Pre- and post-5 week of exercise training period.
  The proportion of participants meeting or exceeding the minimal clinically important difference of ≥1 unit on the Borg 0-10 scale in breathlessness intensity at iso-time of exercise during the cardiopulmonary exercise test (incremental) after the supervised exercise training. A greater score is indicative of worse breathlessness, while a lower score is indicative of lower breathlessness.
Minimal clinically important difference exercise endurance | Pre- and post-5 week of exercise training period.
  The proportion of participants meeting or exceeding the minimal clinically important difference of ≥101-seconds for exercise endurance time at iso-time during the constant-load cardiopulmonary exercise test. The longer the exercise endurance time (greater seconds or minutes) is indicative of a greater improvement in cardiovascular fitness.
Modified Medical Research Council Dyspnea Scale (mMRC) | Pre- and post-5 week of exercise training period.
  The mMRC dyspnea scale will be used to assess change in daily breathlessness pre to post supervised exercise training program. The mMRC dyspnea scale is scored from 0 to 4, where a higher score is indicative of worse daily breathlessness and a lower score is indicative of less daily breathlessness.
COPD Assessment Test | Pre- and post-5 week of exercise training period.
  The COPD Assessment (CAT) Test is a validated test in chronic obstructive pulmonary disease and interstitial lung disease to assess pulmonary and extra-pulmonary symptom burden. The CAT Test will assess changes in pulmonary and extra-pulmonary symptom burden.
Baseline Dyspnea Index and Transition Dyspnea Index | Pre- and post-5 week of exercise training period.
  The Baseline Dyspnea Index (BDI) and Transition Dyspnea Index (TDI) assesses breathlessness burden before and after an intervention or a certain period of time.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Jensen, PhD, Principal Investigator — McGill University
Locations (1):
- Centre of Innovative Medicine of the McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to Dr. Dennis Jensen's Clinical Exercise and Respiratory Physiology Laboratory page — https://www.mcgill.ca/cerpl/